CLINICAL TRIAL: NCT06954129
Title: Markers of Nephrotoxicity During Treatment With Antibiotic Combinations: A Pragmatic Clinical Trial
Brief Title: A Pragmatic Clinical Trial Comparing the Risk of Acute Kidney Injury During Treatment With Vancomycin and Piperacillin-Tazobactam vs. Vancomycin and Cefepime in Hospitalized Patients
Acronym: MONACO
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Todd Miano, Assistant Professor of Epidemiology, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 858301
Record Dates: First submitted 2025-04-23; First posted 2025-05-01 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Acute Kidney Injury
Keywords: vancomycin; piperacillin-tazobactam; cefepime; acute kidney injury; nephrotoxicity; cystatin c; kidney injury molecule 1 (KIM1)
MeSH Terms: conditions — Acute Kidney Injury | interventions — Vancomycin; Piperacillin, Tazobactam Drug Combination; Cefepime

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vancomycin with Piperacillin-Tazobactam (Active Comparator): Participants in the Vancomycin with Piperacillin-Tazobactam arm will be randomized to initial treatment with Vancomycin with Piperacillin-Tazobactam. Subsequent management of antimicrobial treatment will be at the discretion of treating clinicians
  Interventions: Drug: Vancomycin; Drug: Piperacillin-tazobactam
- Vancomycin with Cefepime (Active Comparator): Participants in the Vancomycin with Cefepime arm will be randomized to initial treatment with Vancomycin with Cefepime. Subsequent management of antimicrobial treatment will be at the discretion of treating clinicians
  Interventions: Drug: Vancomycin; Drug: Cefepime

INTERVENTIONS:
Drug: Vancomycin — Vancomycin is a glycopeptide antibiotic used to treat infections caused by Gram-positive bacteria, including those due to methicillin-resistant Staphylococcus aureus. Dosing of vancomycin will follow standard of care procedures, including the use of individualized dosing regimens developed in consultation with clinical pharmacists, based on participant body weight and renal function, and dosage titration guided by therapeutic drug monitoring. Vancomycin is administered via intermittent intravenous infusions of 60-90 minutes.
Drug: Piperacillin-tazobactam — Piperacillin-tazobactam is an anti-pseudomonal penicillin with a dose range of 2.25 g or 4.5 g and frequency of every 6 or 8 hours based on a participant's body weight, renal function, and clinician discretion. Piperacillin-tazobactam is administered via extended-duration (4 hours) intravenous infusions
  Arms: Vancomycin with Piperacillin-Tazobactam
Drug: Cefepime — Cefepime is an anti-pseudomonal cephalosporin with a dose range of 500 mg, 1,000 mg, or 2,000 mg, and frequency every 8, 12, or 24 hours based on a participant's body weight, renal function, and clinician discretion. Cefepime is administered via extended-duration (4 hours) intravenous infusions
  Arms: Vancomycin with Cefepime

SUMMARY:
Hospitalized patients with suspected or confirmed infection are commonly treated with vancomycin (VN) in combination with either piperacillin-tazobactam (PT) or cefepime (CP). Although these regimens have similar effectiveness, recent observational evidence suggests they may differ in terms of the risk for acute kidney injury (AKI). Interpretation of existing evidence is complicated by the limitations of creatinine, the standard biomarker used to monitor kidney function, which has poor sensitivity and specificity for drug induced AKI. To address this important knowledge gap, the investigators propose to conduct a pragmatic, open-label, non-inferiority trial that will examine the comparative risk of AKI between these standard-of-care antibiotic combinations using sensitive and specific markers of drug-induced AKI. We hypothesize that the regimen of VN in combination with PT (VN+PT) is noninferior to the regimen of VN in combination with CP (VN+CP) in terms of AKI risk.

ELIGIBILITY:
Inclusion Criteria:

1. Age of at least 18 years
2. Suspected or confirmed infection based on clinical criteria, for which vancomycin with piperacillin-tazobactam or vancomycin with cefepime was prescribed by the treating clinician, as evidenced by orders being placed in the electronic health record
3. The treating clinician considers both vancomycin with piperacillin- tazobactam or vancomycin with cefepime as acceptable treatment
4. The treating clinician anticipates at least 48 hours of antibiotic treatment

Exclusion Criteria:

1. Dialysis dependence or documented end stage kidney disease
2. AKI at baseline
3. Expected survival <24 hours and/or presence of do not resuscitate orders
4. History of antibiotic-resistant organisms (microbiological culture results showing bacterial isolates with resistant or intermediate susceptibility to any study drug within the prior 90 days)
5. Documented allergy to vancomycin, cephalosporins, or penicillin
6. Suspected central nervous system infection
7. Inability to provide informed consent or lack of proxy for consent
8. Prisoners/incarcerated individuals
9. Known pregnancy or breastfeeding
10. Previous enrollment in this study
11. Receipt of vancomycin, piperacillin-tazobactam, or cefepime for >24 hours within the preceding 7 days. At the time of screening, one-time doses of vancomycin, with or without piperacillin-tazobactam, or cefepime, will be allowed prior to randomization to avoid treatment delays; such patients must be enrolled within twelve hours of antibiotic administration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2029-05 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
Serum Cystatin C Concentration | 5 days post enrollment
  Change in serum cystatin c concentration through Day 5 after antibiotic initiation.

SECONDARY OUTCOMES:
Kidney injury molecule 1 (KIM1) | 5 days post enrollment
  Changes in urinary KIM1 concentration through Day 5 after antibiotic initiation.
Serum creatinine concentration | 5 days post enrollment
  Change in serum creatinine concentration through Day 5 after antibiotic initiation.
Acute Kidney Injury | At 7 and 14 days
  Acute kidney injury as defined by Kidney Disease: Improving Global Outcomes (KDIGO) creatinine criteria:
  Stage 1 AKI (Creatinine increase by 1.5-1.9 times baseline OR increase by >= 0.3 mg/dL) Stage 2 AKI (Creatinine increase by 2.0-2.9 times baseline) Stage 3 AKI (Creatinine increase by >= 3.0 times baseline OR increase to >= 4.0 mg/dL OR New renal replacement therapy (RRT))
Major Adverse Kidney Events (MAKE) | 30 and 60 days
  MAKE consists of death, need for RRT, or persistent kidney dysfunction (decrease in estimated glomerular filtration rate (GFR) to <75% of baseline)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Vaidya VS, Ozer JS, Dieterle F, Collings FB, Ramirez V, Troth S, Muniappa N, Thudium D, Gerhold D, Holder DJ, Bobadilla NA, Marrer E, Perentes E, Cordier A, Vonderscher J, Maurer G, Goering PL, Sistare FD, Bonventre JV. Kidney injury molecule-1 outperforms traditional biomarkers of kidney injury in preclinical biomarker qualification studies. Nat Biotechnol. 2010 May;28(5):478-85. doi: 10.1038/nbt.1623. PMID 20458318
- [Background] Herget-Rosenthal S, Marggraf G, Husing J, Goring F, Pietruck F, Janssen O, Philipp T, Kribben A. Early detection of acute renal failure by serum cystatin C. Kidney Int. 2004 Sep;66(3):1115-22. doi: 10.1111/j.1523-1755.2004.00861.x. PMID 15327406
- [Background] Nejat M, Pickering JW, Walker RJ, Endre ZH. Rapid detection of acute kidney injury by plasma cystatin C in the intensive care unit. Nephrol Dial Transplant. 2010 Oct;25(10):3283-9. doi: 10.1093/ndt/gfq176. Epub 2010 Mar 28. PMID 20350927
- [Background] Bellos I, Karageorgiou V, Pergialiotis V, Perrea DN. Acute kidney injury following the concurrent administration of antipseudomonal beta-lactams and vancomycin: a network meta-analysis. Clin Microbiol Infect. 2020 Jun;26(6):696-705. doi: 10.1016/j.cmi.2020.03.019. Epub 2020 Mar 25. PMID 32222460
- [Background] Pais GM, Liu J, Avedissian SN, Hiner D, Xanthos T, Chalkias A, d'Aloja E, Locci E, Gilchrist A, Prozialeck WC, Rhodes NJ, Lodise TP, Fitzgerald JC, Downes KJ, Zuppa AF, Scheetz MH. Lack of synergistic nephrotoxicity between vancomycin and piperacillin/tazobactam in a rat model and a confirmatory cellular model. J Antimicrob Chemother. 2020 May 1;75(5):1228-1236. doi: 10.1093/jac/dkz563. PMID 32011685
- [Background] Avedissian SN, Pais GM, Liu J, Rhodes NJ, Scheetz MH. Piperacillin-Tazobactam Added to Vancomycin Increases Risk for Acute Kidney Injury: Fact or Fiction? Clin Infect Dis. 2020 Jul 11;71(2):426-432. doi: 10.1093/cid/ciz1189. PMID 31833540
- [Background] Qian ET, Casey JD, Wright A, Wang L, Shotwell MS, Siemann JK, Dear ML, Stollings JL, Lloyd BD, Marvi TK, Seitz KP, Nelson GE, Wright PW, Siew ED, Dennis BM, Wrenn JO, Andereck JW, Han JH, Self WH, Semler MW, Rice TW; Vanderbilt Center for Learning Healthcare and the Pragmatic Critical Care Research Group. Cefepime vs Piperacillin-Tazobactam in Adults Hospitalized With Acute Infection: The ACORN Randomized Clinical Trial. JAMA. 2023 Oct 24;330(16):1557-1567. doi: 10.1001/jama.2023.20583. PMID 37837651
- [Background] Miano TA, Hennessy S, Yang W, Dunn TG, Weisman AR, Oniyide O, Agyekum RS, Turner AP, Ittner CAG, Anderson BJ, Wilson FP, Townsend R, Reilly JP, Giannini HM, Cosgriff CV, Jones TK, Meyer NJ, Shashaty MGS. Association of vancomycin plus piperacillin-tazobactam with early changes in creatinine versus cystatin C in critically ill adults: a prospective cohort study. Intensive Care Med. 2022 Sep;48(9):1144-1155. doi: 10.1007/s00134-022-06811-0. Epub 2022 Jul 14. PMID 35833959
- [Background] Rhodes A, Evans LE, Alhazzani W, Levy MM, Antonelli M, Ferrer R, Kumar A, Sevransky JE, Sprung CL, Nunnally ME, Rochwerg B, Rubenfeld GD, Angus DC, Annane D, Beale RJ, Bellinghan GJ, Bernard GR, Chiche JD, Coopersmith C, De Backer DP, French CJ, Fujishima S, Gerlach H, Hidalgo JL, Hollenberg SM, Jones AE, Karnad DR, Kleinpell RM, Koh Y, Lisboa TC, Machado FR, Marini JJ, Marshall JC, Mazuski JE, McIntyre LA, McLean AS, Mehta S, Moreno RP, Myburgh J, Navalesi P, Nishida O, Osborn TM, Perner A, Plunkett CM, Ranieri M, Schorr CA, Seckel MA, Seymour CW, Shieh L, Shukri KA, Simpson SQ, Singer M, Thompson BT, Townsend SR, Van der Poll T, Vincent JL, Wiersinga WJ, Zimmerman JL, Dellinger RP. Surviving Sepsis Campaign: International Guidelines for Management of Sepsis and Septic Shock: 2016. Intensive Care Med. 2017 Mar;43(3):304-377. doi: 10.1007/s00134-017-4683-6. Epub 2017 Jan 18. PMID 28101605
- [Background] Cecconi M, Evans L, Levy M, Rhodes A. Sepsis and septic shock. Lancet. 2018 Jul 7;392(10141):75-87. doi: 10.1016/S0140-6736(18)30696-2. Epub 2018 Jun 21. PMID 29937192